CLINICAL TRIAL: NCT05451732
Title: New Autologous Fat Graft for the Treatment of Urethral Stricture
Brief Title: Nanofat Grafting in Male and Female Subjects Affected by Urethral Strictures
Acronym: NFUS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Roma La Sapienza (Other)
Collaborators: University of Pisa (Other)
Responsible Party: Principal Investigator, Antonio Luigi Pastore, Associate Professor, University of Roma La Sapienza
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Urethral Strict and Naofat
Record Dates: First submitted 2022-04-04; First posted 2022-07-11 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-07

CONDITIONS: Urethral Stricture
MeSH Terms: conditions — Urethral Stricture

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nanofat grafting (Experimental): Nanofat grafting with tissue transfer by injection in the urethral stricture
  Interventions: Procedure: Nanofat grafting

INTERVENTIONS:
Procedure: Nanofat grafting — Naofat grafting in the urethral stricture. The autologous adipose tissue is transferred by injection and in this way, the access to the urethral stricture is carried out with a minimal incision of the male urethra while in the female urethra is transferred exclusively with injections, without incision of urethral tissue.

SUMMARY:
In 2001 Zuk showed that lipoaspirate contains multipotent adipose stem cells (ADSCs) like in the bone marrow, thereby expanding opportunities in multiple fields. ADSCs have emerged as a key element of regenerative medicine surgery due to their ability to differentiate into a variety of different cell lineages. Moreover, their capacity of paracrine secretion of a broad selection of cytokines, chemokines, and growth factors makes them highly clinically attractive. More specific, of particular interest are the anti-apoptotic, anti-inflammatory, proangiogenic, immunomodulatory, and anti-scarring effects that have been demonstrated for ADSCs, which effects on wound healing, soft-tissue restoration, and scar remodeling.

Nanofat firstly introduced by Tonnard in 2013, is an ultra-purified adipose tissue-derived product that is devoid of mature adipocytes but rich in ADSCs and with regenerative properties.

Nanofat represents a particular formulation of adipose grafting because it is liquid and it is easily transferable to tissues by injection. The nanofat because is free of whole adipocytes does not have the side effects of others adipose-derived formulations containing whole adipocytes (microfat, lipofilling, macrofat), such as the formation of deposits, granulomas, oily cysts, keloids.

Investigators aim to evaluate the use of nanofat grafting in the treatment in urethral strictures of the female and male urethras.

DETAILED DESCRIPTION:
Urethral stricture is the reduction of the urethral lumen due to the growth of scar tissue inside the urethral wall, due to various causes.

In the last thirty years, in reconstructive urethral surgery have been described several urethroplasties to repair the urethra and to restore urinary flow.

Obstructed stricture were treated with the removal of the urethral tract stricture and with the anastomosis of the two urethral stumps by the technique called "end-to end anastomosis". This technique is today reserved only for cases of complete urethral stricture of the male urethra because it causes many negative consequences on the sexual activity: shortening of the urethra and the penis, abnormal curvature of the penis in erection, reduction of penile sensitivity. In female urethral stricture this technique has never been used.

Many urethroplasties have been described with the enlargement of the urethra with a good success rate, but some risks such as the formation of fistulas and redo of the stricture. Today several autologous graft tissues are used including the genital and extragenital skin and the buccal mucosa. The use of preputial skin requires complete circumcision and is often not accepted by the patient. The use of extragenital skin is invasive and is used in some long male urethral stricture, while it is not used in female urethral reconstruction.

The buccal mucosa is today considered the optimal graft tissue, due to its histological characteristics that make it suitable for the reparative urethral surgery. However, it must be considered that the withdrawal can be a potential cause of oral complications and, moreover, there is a limit to the length of the tissue that can be taken and is a medium invasive procedure, with discomfort of the patient in the days following the harvest.

Over the last decade, many tissue engineering have been carried out in an attempt to create a tissue that could have the appropriate histological characteristics and size, but without the risk of complications related to the harvest. Many studies have concluded that tissue engineering is not usable except in specialized laboratories, because of its high costs and because not given satisfactory results.

Since 2001, the new concept of "tissue regeneration" has been born through plastic surgery techniques that involve the use of ultra-purified adipose tissue graft rich in stem cells and growth factors that regenerate scar tissues, as the urethral stricture.

In 2001 Zuk showed that lipoaspirate contains multipotent adipose stem cells (ADSCs) like in the bone marrow, thereby expanding opportunities in multiple fields. ADSCs have emerged as a key element of regenerative medicine surgery due to their ability to differentiate into a variety of different cell lineages. Moreover, their capacity of paracrine secretion of a broad selection of cytokines, chemokines, and growth factors makes them highly clinically attractive. More specific, of particular interest are the anti-apoptotic, anti-inflammatory, proangiogenic, immunomodulatory, and anti-scarring effects that have been demonstrated for ADSCs, which effects on wound healing, soft-tissue restoration, and scar remodeling.

Nanofat firstly introduced by Tonnard in 2013, is an ultra-purified adipose tissue-derived product that is devoid of mature adipocytes but rich in ADSCs and with regenerative properties.

Nanofat represents a particular formulation of adipose grafting because it is liquid and it is easily transferable to tissues by injection. The nanofat because is free of whole adipocytes does not have the side effects of others adipose-derived formulations containing whole adipocytes (microfat, lipofilling, macrofat), such as the formation of deposits, granulomas, oily cysts, keloids.

We aim to investigate the use of nanofat grafting in the treatment in urethral strictures of the female and male urethras.

Broad-spectrum antibiotic prophylaxis amoxicillin + clavulanic acid is carried out one hour before anesthesia.

After infiltration procedure with Klein's solution in the donor area, the lipoaspirate was obtained by means of a small 3 mm multiport collection cannula with 1 mm diameter side holes. The collection cannula was connected to a 60 ml syringe and the syringe plunger was pulled back to create an adequate negative pressure. The adipose tissue was decanted. At the end of liposuction, the contour deformities of the donor area were prevented by using a smaller diameter cannula, avoiding aspirations from the superficial layers, employing a "crossing" technique and allowing a slight under correction.

To obtain the nanofat, according to Tonnard's technique, the emulsification was obtained by moving the fat between two 10 cc syringes connected by a 1.4 mm connector. The same procedure is repeated with a 1.2 mm connector. This progressive emulsification process is important to ensure the destruction of all adipocytes. The product is then passed through a 400- or 600-micron filter to remove the connective tissue. In this way the liposuction become into nanofat. The nanofat in a 10-cc syringe connected with a 25 gauge needle is then used to create tunnels in the plane of the sclerotic tissues and the nanofat is introduced into the tunnels. Unlike other autologous grafts (skin and mucous membranes) the adipose tissue is transferred by injection and in this way access to urethral stricture is carried out with a minimal incision of the male urethra while in the female urethra is transferred exclusively with injections, without incision of urethral or genital tissue.

A catheter is left in place for 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Urethral stricture naive or recurrent in male and female patients aged > 18 y.o.

Exclusion Criteria:

* Neurogenic urinary tract disorders
* Urinary tract infections
* Age < 18 y.o.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-12-15 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
uroflow time 1 | 90 days after nonfat grafting
  Uroflowmetry examination (ml/sec)
uroflow time 2 | 180 days after nonfat grafting
  Uroflowmetry examination (ml/sec)
Functional time 1 | 90 days after nonfat grafting
  Post ovoidal residue (ML)
Functional time 2 | 180 days after nonfat grafting
  Post ovoidal residue (ML)

CONTACTS AND LOCATIONS:
Locations (1):
- Antonio Luigi Pastore, Latina, Italy

IPD SHARING:
Plan to Share IPD: Yes
All IPD will be shared with other researchers
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Every 4 weeks
Access Criteria: by mail

REFERENCES:
- [Background] Tonnard P, Verpaele A, Peeters G, Hamdi M, Cornelissen M, Declercq H. Nanofat grafting: basic research and clinical applications. Plast Reconstr Surg. 2013 Oct;132(4):1017-1026. doi: 10.1097/PRS.0b013e31829fe1b0. PMID 23783059